CLINICAL TRIAL: NCT00838539
Title: A Phase 1 Study Of Neratinib In Combination With Temsirolimus In Subjects With Solid Tumors
Brief Title: Study Evaluating Neratinib In Combination With Temsirolimus In Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Puma Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3144A1-2205 / B1891016
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-08

CONDITIONS: Neoplasms; Malignant Carcinoma
Keywords: Neratinib; solid tumors; phase 1; dose finding study; HKI-272; Nerlynx; Temsirolimus; PB-272
MeSH Terms: conditions — Neoplasms | interventions — neratinib; temsirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- Neratinib and Temsirolimus (Dose level 1) (Experimental): Neratinib 120 mg and Temsirolimus 15 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 2) (Experimental): Neratinib 120 mg and Temsirolimus 25 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 3) (Experimental): Neratinib 120 mg and Temsirolimus 50 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 4) (Experimental): Neratinib 120 mg and Temsirolimus 75 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 5) (Experimental): Neratinib 160 mg and Temsirolimus 15 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 6) (Experimental): Neratinib 160 mg and Temsirolimus 25 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 7) (Experimental): Neratinib 160 mg and Temsirolimus 50 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 8) (Experimental): Neratinib 160 mg and Temsirolimus 75 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 9) (Experimental): Neratinib 200 mg and Temsirolimus 15 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 10) (Experimental): Neratinib 200 mg and Temsirolimus 25 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 11) (Experimental): Neratinib 200 mg and Temsirolimus 50 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus
- Neratinib and Temsirolimus (Dose level 12) (Experimental): Neratinib 240 mg and Temsirolimus 15 mg: Neratinib 40 mg tablets administered orally daily for as long as tolerated and the disease under study does not worsen. Temsirolimus administered intravenously once weekly for as long as tolerated and the disease under study does not worsen
  Interventions: Drug: Neratinib; Drug: Temsirolimus

INTERVENTIONS:
Drug: Neratinib
  Other Names: HKI-272
Drug: Temsirolimus
  Other Names: Torisel, CCI-779

SUMMARY:
The primary purpose of this study is to identify the maximum tolerated dose(s) (MTD) of neratinib in combination with temsirolimus in subjects with solid tumors. This study will also include a preliminary evaluation of efficacy, and assessment of pharmacokinetic (PK) parameters of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of advanced or metastatic solid tumor.
* Measurable disease per Response Criteria in Solid Tumors (RECIST criteria).
* Incurable cancer, with disease progression following at least 1 conventional or standard therapy for locally advanced or metastatic disease.
* Negative pregnancy test for women of child bearing potential.

Exclusion Criteria:

* Chronic treatment with corticosteroids.
* Primary central nervous system (CNS) tumors and active metastases.
* Presence of clinically significant or uncontrolled cardiac disease.
* Significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom.
* Symptomatic or prior history of non-infectious interstitial pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puma, Study Director — Biotechnology
Locations (4):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
- Institut Gustave Roussy, Villejuif, France

REFERENCES:
- [Derived] Gandhi L, Bahleda R, Tolaney SM, Kwak EL, Cleary JM, Pandya SS, Hollebecque A, Abbas R, Ananthakrishnan R, Berkenblit A, Krygowski M, Liang Y, Turnbull KW, Shapiro GI, Soria JC. Phase I study of neratinib in combination with temsirolimus in patients with human epidermal growth factor receptor 2-dependent and other solid tumors. J Clin Oncol. 2014 Jan 10;32(2):68-75. doi: 10.1200/JCO.2012.47.2787. Epub 2013 Dec 9. PMID 24323026

RESULTS

PARTICIPANT FLOW:
Groups:
- N120 + T15: Neratinib 120 mg + Temsirolimus 15 mg
- N120 + T25: Neratinib 120 mg + Temsirolimus 25 mg
- N120 + T50: Neratinib 120 mg + Temsirolimus 50 mg
- N120 + T75: Neratinib 120 mg + Temsirolimus 75 mg
- N160 + T15: Neratinib 160 mg + Temsirolimus 15 mg
- N160 + T25: Neratinib 160 mg + Temsirolimus 25 mg
- N160 + T50: Neratinib 160 mg + Temsirolimus 50 mg
- N160 + T75: Neratinib 160 mg + Temsirolimus 75 mg
- N200 + T15: Neratinib 200 mg + Temsirolimus 15 mg
- N200 + T25: Neratinib 200 mg + Temsirolimus 25 mg
- N200 + T50: Neratinib 200 mg + Temsirolimus 50 mg
- N240 + T15: Neratinib 240 mg + Temsirolimus 15 mg
Period: Overall Study
Arm/Group | N120 + T15 | N120 + T25 | N120 + T50 | N120 + T75 | N160 + T15 | N160 + T25 | N160 + T50 | N160 + T75 | N200 + T15 | N200 + T25 | N200 + T50 | N240 + T15
Started | 3 | 6 | 5 | 4 | 6 | 4 | 7 | 6 | 5 | 8 | 5 | 4
Received Treatment | 3 | 5 | 5 | 4 | 4 | 4 | 7 | 6 | 5 | 8 | 5 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 6 | 5 | 4 | 6 | 4 | 5 | 6 | 5 | 8 | 5 | 4
Not completed — Disease Progression | 2 | 4 | 3 | 2 | 4 | 2 | 3 | 4 | 4 | 5 | 1 | 4
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 2 | 0 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Clinical Progression | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- N120 + T15: Neratinib 120 mg qd + Temsirolimus 15 mg, IV, weekly
- N120 + T25: Neratinib 120 mg qd + Temsirolimus 25 mg, IV, weekly
- N120 + T50: Neratinib 120 mg qd + Temsirolimus 50 mg, IV, weekly
- N120 + T75: Neratinib 120 mg qd + Temsirolimus 75mg, IV, weekly
- N160 + T15: Neratinib 160 mg qd + Temsirolimus 15 mg, IV, weekly
- N160 + T25: Neratinib 160 mg qd + Temsirolimus 25 mg, IV, weekly
- N160 + T50: Neratinib 160 mg qd + Temsirolimus 50 mg, IV, weekly
- N160 + T75: Neratinib 160 mg qd + Temsirolimus 75 mg, IV, weekly
- N200 + T15: Neratinib 200 mg qd + Temsirolimus 15 mg, IV, weekly
- N200 + T25: Neratinib 200 mg qd + Temsirolimus 25 mg, IV, weekly
- N200 + T50: Neratinib 200 mg qd + Temsirolimus 50 mg, IV, weekly
- N240 + T15: Neratinib 240 mg qd + Temsirolimus 15 mg, IV, weekly
- Total: Total of all reporting groups
Arm/Group | N120 + T15 | N120 + T25 | N120 + T50 | N120 + T75 | N160 + T15 | N160 + T25 | N160 + T50 | N160 + T75 | N200 + T15 | N200 + T25 | N200 + T50 | N240 + T15 | Total
Number analyzed (Participants) | 3 | 5 | 5 | 4 | 4 | 4 | 7 | 6 | 5 | 8 | 5 | 4 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 4 | 4 | 4 | 4 | 4 | 6 | 5 | 3 | 7 | 5 | 4 | 52
  >=65 years | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.00 (26.15) | 58.60 (10.26) | 43.00 (16.40) | 49.50 (7.94) | 49.75 (4.79) | 49.75 (5.68) | 49.29 (12.20) | 53.17 (11.62) | 59.60 (10.62) | 44.50 (18.72) | 50.00 (7.00) | 56.75 (5.74) | 50.82 (12.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 1 | 4 | 3 | 4 | 4 | 5 | 4 | 3 | 4 | 4 | 40
  Male | 2 | 2 | 4 | 0 | 1 | 0 | 3 | 1 | 1 | 5 | 1 | 0 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race was not reported for 31 subjects in site in France.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
    White | 1 | 3 | 2 | 1 | 1 | 3 | 4 | 3 | 2 | 2 | 3 | 1 | 26
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 2 | 2 | 3 | 3 | 3 | 1 | 3 | 3 | 3 | 5 | 1 | 2 | 31

OUTCOME MEASURES:

1. Primary Outcome: Probability of Dose-Limiting Toxicity (DLT)
Description: A DLT was defined as any dose-limiting Adverse Event related to neratinib + Temsirolimus as Grade 3 or higher nonhematologic toxicity (except neutropenia) or Grade 3 or higher diarrhea lasting >2 days with optimal antidiarrheal therapy etc.
Time Frame: From first dose date to day 28
Population: Evaluable subjects for the Maximum Tolerated Dose (MTD) contour estimation were those who either experienced a DLT within the first 28 days, regardless of the number of doses of treatment received, or received at least 21 doses of neratinib and at least 2 doses of Temsirolimus in the first 28 days of treatment.
Measure: Number; unit: percent probability
Groups:
- Neratinib 120 mg: Neratinib 120 mg/day with indicated level of Temsirolimus, weekly, IV.
- Neratinib 160 mg: Neratinib 160 mg/day with indicated level of Temsirolimus, weekly, IV.
- Neratinib 200 mg: Neratinib 200 mg/day with indicated level of Temsirolimus, weekly, IV.
- Neratinib 240 mg: Neratinib 240 mg/day with indicated level of Temsirolimus, weekly, IV.
Arm/Group | Neratinib 120 mg | Neratinib 160 mg | Neratinib 200 mg | Neratinib 240 mg
Number analyzed (Participants) | 14 | 20 | 13 | 4
percent probability
  Temsirolimus 15 mg: number analyzed (Participants) | 2 | 4 | 4 | 4
  Temsirolimus 15 mg | 0 | 12.5 | 12.5 | 50
  Temsirolimus 25 mg: number analyzed (Participants) | 4 | 4 | 8 | 0
  Temsirolimus 25 mg | 13.63 | 13.64 | 12.5 |
  Temsirolimus 50 mg: number analyzed (Participants) | 4 | 6 | 1 | 0
  Temsirolimus 50 mg | 13.63 | 13.64 | 100 |
  Temsirolimus 75 mg: number analyzed (Participants) | 4 | 6 | 0 | 0
  Temsirolimus 75 mg | 13.63 | 50 |  |

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Neratinib in Combination With Temsirolimus
Description: Identification of the daily neratinib high-dose MTD in combination with weekly temsirolimus.
Time Frame: From first dose date to day 28
Population: Evaluable subjects were those that either experienced a dose limiting toxicity within the first 28 days, regardless of the number of doses of treatment received, or those that received at least 21 doses of neratinib and at least 2 doses of Temsirolimus in the first 28 days of treatment at the original dose level prescribed.
Measure: Number; unit: mg
Groups:
- MTD Ner With TEMS: Neratinib MTD in combination with Temsirolimus
Arm/Group | MTD Ner With TEMS
Number analyzed (Participants) | 51
mg | 200

3. Primary Outcome: Maximum Tolerated Dose (MTD) of Temsirolimus in Combination With Neratinib
Description: Identification of the weekly temsirolimus high-dose MTD in combination with daily neratinib
Time Frame: From first dose date to day 28
Population: Evaluable subjects include those that either experienced a dose limiting toxicity within the first 28 days, regardless of the number of doses of treatment received, or those that received at least 21 doses of neratinib and at least 2 doses of Temsirolimus in the first 28 days of treatment at the original dose level prescribed.
Measure: Number; unit: mg
Groups:
- MTD TEMS With Ner: Temsirolimus MTD in combination with Neratinib
Arm/Group | MTD TEMS With Ner
Number analyzed (Participants) | 51
mg | 50

4. Primary Outcome: Adverse Events Causing Dose Limiting Toxicities
Description: A DLT was defined as any dose-limiting adverse event (AE) related to neratinib + TEMSR as follows: [1] Grade 3 or 4 nonhematologic toxicity (Grade 3 or 4 nausea, vomiting, hyperglycemia, hypophosphatemia, hypertriglyceridemia, or hypercholesterolemia was not considered a DLT unless the subject was already receiving optimal medical therapy). [2] Grade 3 or 4 diarrhea lasting >2 days while subject was on optimal vigorous antidiarrheal therapy.
  [3] Grade 4 neutropenia lasting >3 days or Grade 3 or 4 neutropenia of any duration with sepsis or a fever >38.5C. [4] Platelet value less than or equal to 25,000/mm3 or bleeding requiring a platelet transfusion. [5] Delayed recovery from toxicity, which delayed rescheduled re-treatment for >3 weeks. [6] Inability to maintain the original dose during the first 28 days of treatment (at least 21 doses of neratinib and 2 doses of TEMSR at the original specified dose) due to treatment-related toxicity.
Time Frame: From first dose date to day 21
Measure: Count of Participants; unit: Participants
Arm/Group | N120 + T15 | N120 + T25 | N120 + T50 | N120 + T75 | N160 + T15 | N160 + T25 | N160 + T50 | N160 + T75 | N200 + T15 | N200 + T25 | N200 + T50 | N240 + T15
Number analyzed (Participants) | 3 | 5 | 5 | 4 | 4 | 4 | 7 | 6 | 5 | 8 | 5 | 4
Participants | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 1 | 1 | 2

5. Secondary Outcome: Best Overall Response
Description: The best overall response was described using the data as reported by study center investigators per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first dose date to progression/death or last tumor assessment, up to 30 months
Population: Subjects who completed at least 1 tumor assessment post-baseline after starting treatment and received sufficient drug (>= 21 doses of neratinib and >= 2 doses of temsirolimus in the first 28 days unless the subject discontinued treatment early for documented progression or symptomatic deterioration after taking at least 1 dose of test article[s])
Measure: Count of Participants; unit: Participants
Groups:
- Neratinib 120 mg + Temsirolimus: Neratinib 120 mg, qd, with various dose levels of temsirolimus, IV, once weekly.
- Neratinib 160 mg + Temsirolimus: Neratinib 160 mg, qd, with various dose levels of temsirolimus, IV, once weekly.
- Neratinib 200 mg + Temsirolimus: Neratinib 200 mg, qd, with various dose levels of temsirolimus, IV, once weekly.
- Neratinib 240 mg + Temsirolimus: Neratinib 240 mg, qd, with various dose levels of temsirolimus, IV, once weekly.
Arm/Group | Neratinib 120 mg + Temsirolimus | Neratinib 160 mg + Temsirolimus | Neratinib 200 mg + Temsirolimus | Neratinib 240 mg + Temsirolimus
Number analyzed (Participants) | 13 | 18 | 10 | 4
Participants
  Complete Response | 1 | 0 | 1 | 0
  Partial Response | 1 | 3 | 1 | 1
  Stable Disease | 8 | 11 | 6 | 1
  Progressive Disease | 3 | 3 | 2 | 1
  Unknown | 0 | 1 | 0 | 1

6. Secondary Outcome: Clinical Benefit Rate
Description: Percentage of subjects with a complete response, partial response, or stable disease >= 24 weeks, as determined by investigator assessment per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first dose date to progression/death or last tumor assessment, up to 30 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib 120 mg + Temsirolimus | Neratinib 160 mg + Temsirolimus | Neratinib 200 mg + Temsirolimus | Neratinib 240 mg + Temsirolimus
Number analyzed (Participants) | 13 | 18 | 10 | 4
percentage of participants | 38.5 [13.86 to 68.42] | 27.8 [9.69 to 53.48] | 20.0 [2.52 to 55.61] | 25.0 [0.63 to 80.59]

7. Secondary Outcome: Objective Response Rate
Description: Percentage of subjects with a complete response (CR) or partial response (PR) per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR. Progression is defined as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: From first dose date to progression/death or last tumor assessment, up to 30 months
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Neratinib 120 mg + Temsirolimus | Neratinib 160 mg + Temsirolimus | Neratinib 200 mg + Temsirolimus | Neratinib 240 mg + Temsirolimus
Number analyzed (Participants) | 13 | 18 | 10 | 4
percentage of participants | 15.4 [1.92 to 45.45] | 16.7 [3.58 to 41.42] | 20.0 [2.52 to 55.61] | 25.0 [0.63 to 80.59]

8. Secondary Outcome: Area Under the Curve Tau
Description: Area Under the Curve tau of neratinib concentrations, collected at 2, 4, 8, and 24 hours post-neratinib administration, at the week 4 dose.
Time Frame: Week 4
Population: Subjects who had pharmacokinetic concentrations available at the dose combination, at day 22.
Measure: Geometric Mean (Full Range); unit: ng*hr/mL
Groups:
- Temsirolimus 15 mg; Temsirolimus 25 mg: Neratinib at indicated dose levels with Temsirolimus 15 mg, IV, once weekly
- Temsirolimus 50 mg: Neratinib at indicated dose levels with Temsirolimus 50 mg, IV, once weekly
- Temsirolums 75 mg: Neratinib at indicated dose levels with Temsirolimus 75 mg, IV, once weekly
Arm/Group | Temsirolimus 15 mg | Temsirolimus 25 mg | Temsirolimus 50 mg | Temsirolums 75 mg
Number analyzed (Participants) | 11 | 15 | 11 | 9
ng*hr/mL
  Neratinib 120 mg | 390.65 [181.99 to 838.56] | 621.20 [295.20 to 1836.82] | 408.98 [45.61 to 1034.19] | 477.37 [188.73 to 1036.40]
  Neratinib 160 mg | 1146.53 [557.94 to 2356.03] | 775.89 [590.90 to 1232.98] | 640.36 [378.53 to 1617.55] | 753.47 [323.88 to 1486.12]
  Neratinib 200 mg | 1396.48 [627.10 to 2256.55] | 357.30 [33.16 to 790.08] | 963.19 [963.19 to 963.19] | NA [NA to NA] — Dose combination not studied
  Neratinib 240 mg | 1402.37 [519.81 to 2602.27] | NA [NA to NA] — Dose combination not studied | NA [NA to NA] — Dose combination not studied | NA [NA to NA] — Dose combination not studied

ADVERSE EVENTS:
Time Frame: From first dose through 28 days after last dose, up to 30 months.
Groups:
- N120 + T75: Neratinib 120 mg qd + Temsirolimus 75 mg, IV, weekly
Arm/Group | N120 + T15 | N120 + T25 | N120 + T50 | N120 + T75 | N160 + T15 | N160 + T25 | N160 + T50 | N160 + T75 | N200 + T15 | N200 + T25 | N200 + T50 | N240 + T15
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/6 | 1/5 | 1/4 | 3/6 | 2/4 | 5/7 | 3/6 | 4/5 | 5/8 | 3/5 | 3/4
Other Adverse Events (participants affected / at risk) | 3/3 | 5/6 | 5/5 | 4/4 | 4/6 | 4/4 | 7/7 | 6/6 | 5/5 | 8/8 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | N120 + T15 (N=3) | N120 + T25 (N=6) | N120 + T50 (N=5) | N120 + T75 (N=4) | N160 + T15 (N=6) | N160 + T25 (N=4) | N160 + T50 (N=7) | N160 + T75 (N=6) | N200 + T15 (N=5) | N200 + T25 (N=8) | N200 + T50 (N=5) | N240 + T15 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lung abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radiculopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | N120 + T15 (N=3) | N120 + T25 (N=6) | N120 + T50 (N=5) | N120 + T75 (N=4) | N160 + T15 (N=6) | N160 + T25 (N=4) | N160 + T50 (N=7) | N160 + T75 (N=6) | N200 + T15 (N=5) | N200 + T25 (N=8) | N200 + T50 (N=5) | N240 + T15 (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 3 | 3 | 2 | 3 | 3 | 4 | 4 | 2 | 2 | 2 | 3
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 3 | 0 | 1 | 0 | 0 | 2 | 1 | 2 | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 2 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 3 | 2 | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 3 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2 | 2 | 2 | 0 | 1 | 3 | 3 | 3 | 4 | 4 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Ear pruritus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eyelid function disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Keratitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Vitreous floaters (Eye disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2 | 2 | 0 | 0 | 0 | 2 | 0 | 1 | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0
Aerophagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 2 | 2 | 3 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 3 | 1 | 1 | 2 | 1 | 1 | 2 | 2 | 5 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 5 | 5 | 4 | 3 | 4 | 7 | 5 | 5 | 6 | 4 | 4
Distal ileal obstruction syndrome (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 3 | 2 | 3 | 2 | 3 | 5 | 2 | 5 | 4 | 2 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 2 | 3 | 3 | 2 | 2 | 3 | 3 | 2 | 5 | 3 | 2
Subileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 3 | 1 | 3 | 2 | 2 | 5 | 2 | 4 | 4 | 1 | 4
Asthenia (General disorders) | 2 | 2 | 2 | 2 | 3 | 1 | 3 | 3 | 3 | 5 | 1 | 2
Catheter site haemorrhage (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 2 | 0 | 2 | 2 | 4 | 0 | 1 | 2 | 1 | 1
Granuloma (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 3 | 0 | 3 | 2 | 4 | 3 | 2 | 1 | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 3 | 3 | 2 | 3 | 1 | 4 | 0 | 2 | 5 | 1 | 1
Thrombosis in device (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Xerosis (General disorders) | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 1 | 0 | 2 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Botryomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Ecthyma (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipeloid (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Folliculitis (Infections and infestations) | 0 | 1 | 2 | 1 | 3 | 1 | 2 | 3 | 0 | 5 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Lymphangitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 1 | 3 | 1 | 1 | 2 | 1 | 1 | 2 | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 1 | 0 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Vaginal infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis radiation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 3 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 3 | 2 | 1 | 2 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Blood creatine phosphokinase (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0
Cardiac murmur (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest X-ray abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 0 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 2 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 3 | 0 | 3 | 1 | 2 | 5 | 2 | 3 | 3 | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 2 | 2 | 0 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 3 | 2 | 1 | 1 | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 4 | 2 | 2 | 1 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1 | 1 | 2 | 4 | 1 | 2 | 1 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 0 | 0 | 2 | 3 | 2 | 2 | 1 | 1 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2 | 2 | 2 | 3 | 1 | 1 | 3 | 1 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 2 | 0 | 3 | 3 | 2 | 2 | 4 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 6 | 1 | 1 | 4 | 0 | 4
Polydipsia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 3 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 2 | 1 | 3 | 1 | 1 | 1 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tumour embolism (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 1 | 0 | 3 | 0 | 2 | 3 | 2 | 1 | 1 | 0 | 1
Dystonia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 4 | 2 | 2 | 1 | 1 | 1 | 1 | 3 | 4 | 0 | 2
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorgasmia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 1 | 1 | 2 | 2 | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Genital rash (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Penile erythema (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vaginal inflammation (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal lesion (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 1 | 1 | 3 | 1 | 4 | 2 | 0 | 4 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 4 | 2 | 3 | 1 | 0 | 2 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 1 | 2 | 1 | 3 | 3 | 0 | 3 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 2 | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 1 | 0 | 0
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nail toxicity (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 2 | 1 | 2 | 2 | 5 | 1 | 2 | 3 | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 1 | 1 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Xeroderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less